CLINICAL TRIAL: NCT00218205
Title: A Phase II Trial of Epirubicin With Estramustine Phosphate and Celecoxib for the Treatment of Hormone Resistant Prostate Cancer (HRPC)
Brief Title: A Study of Epirubicin With Estramustine Phosphate and Celecoxib for the Treatment of Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Veterans Affairs, New Jersey (U.S. Federal Agency)
Collaborators: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-EPIRU-0030-280-US
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Prostate Cancer
Keywords: Epirubicin; Estramustine Phosphate; Celecoxib; Hormone Refractory Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Epirubicin; Estramustine; Celecoxib

INTERVENTIONS:
Drug: Epirubicin
Drug: Estramustine Phosphate
Drug: Celecoxib

SUMMARY:
The purpose of this clinical trial is to find out the effect of epirubicin with estramustine phosphate and celecoxib on PSA and objective response in patients with hormone resistant prostate cancer as well as evaluating the toxicity, quality of life of this combination. Celecoxib is an FDA approved drug to treat arthritis. Epirubicin, alone or with estramustine phosphate has been used in the treatment of hormone resistant prostate cancer. These drugs have demonstrated evidences of tumor blood vessel suppression and combination of these three drugs could possibly arrest further tumor growth or even make the tumor decrease in size.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically proven adenocarcinoma of the prostate gland.
* Patient must have evidence of progressive metastatic disease (e.g., bone, pelvic mass, lymph node, liver or lung metastases) within 6 weeks prior to participation in the study.
* Patients must not have an elevated PSA level as the only evidence of disease. While castrated, the patients should have rising PSA on two consecutive measurements at least 1 week apart. The confirmatory PSA must be obtained within 1 week prior to study registration and should be >10ng/ml.
* Patients with bone metastases only (i.e., lacking soft-tissue disease) must have a PSA level of > 10 ng/ml. Patients with soft tissue metastases and /or visceral disease must have either measurable disease or a PSA level of > 10 ng/ml.
* Radiological evidence of hydronephrosis will not by itself constitute evidence of metastatic disease.
* Patients must have had prior treatment with bilateral orchiectomy or other primary hormonal therapy (e.g., estrogen therapy, LHRH analog + flutamide, etc.) with evidence of treatment failure.

NOTE: Patients who have not undergone bilateral orchiectomy must continue LHRH agonist therapy (e.g., depot leuprolide or goserelin) while receiving this protocol therapy.

* For patients previously treated with flutamide (Eulexin), nilutamide (Nilandron), or bicalutamide (Casodex): Patients must have discontinued flutamide or nilutamide < 4 weeks and for bicalutamide 6 weeks prior to registration.
* Patients should not have prior exposure to anthracyclines or estramustine phosphate.
* Patients must not have had prior radiotherapy < 4 weeks prior to this protocol treatment.
* Patients must not have previously received Strontium 89, Samarium 153, or other radioisotope therapies.
* Patients must have recovered from all toxicities due to prior treatment for prostate cancer prior to receiving this protocol treatment.
* Patients must have adequate bone marrow function: (WBC > 4000/ mm3, granulocytes > 2000/ mm3, platelet count > 100,000/mm3, and Hemoglobin > 8.0 g/dl < 4 weeks prior to participate in this study.
* Patients must have the following chemistry values < 4 weeks prior to participate in this study:
* Bilirubin < 1.5 mg/dl
* Transaminases (SGOT and/or SGPT) < 5 x institutional upper limit of normal (ULN)
* Creatinine < 2.0 mg/d. or creatinine clearance > 50 ml/min
* Alkaline phosphatase £ 5 x ULN
* Patients must have no active angina pectoris, or known heart disease of New York Heart Association Class III-IV. Patients must not have a history of myocardial infarction < 6 months prior to the study participation.
* Patients with a history of prior malignancy are eligible provided they were treated with curative intent and have been free of disease for the time period considered appropriate for the specific cancer.
* No serious concurrent medical illness or active infection should be present which would jeopardize the ability of the patient to receive the chemotherapy outlined in this protocol with reasonable safety.
* Sexually active patients must use an accepted and effective method of contraception while receiving protocol treatment.
* Patients must have a Karnofsky Performance Scale (KPS) score over 50. (Equaling ECOG Performance Scale of 0, 1, or 2).
* Age > 18 years.
* Patient must have failed the Taxotere treatment.

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2002-07; Study Completion 2006-06

PRIMARY OUTCOMES:
Determine the effect of epirubicin with estramustine phosphate and celecoxib on PSA and objective response in patients with HRPC

SECONDARY OUTCOMES:
Evaluate the toxicity of the combination of epirubicin with estramustine phosphate and celecoxib in patients with stage D3 prostate cancer.
Determine the effects of this regimen on quality of life.
Determine the survival of the patients treated with the proposed regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Basil Kasimis, MD, Principal Investigator — Department of Veterans Affairs NJ Health Care System
Locations (1):
- Department of Veterans Affairs NJ Health Care System, East Orange, New Jersey, United States

REFERENCES:
- [Result] Zhong F, Kasimis B, Hwang S, Cogswell J, Chang V, Morales E, Gonzalez M, Boholli I, Ohanian M, Blumenfrucht M: Second Line Treatment of Hormone Resistant Prostate Cancer (HRPC). A Phase II Trial of Epirubicin (E), Estramustine Phosphate (EP) and Celecoxib © Proc Am Soc Clin Oncol, Vol 24 #4754, 2005.